CLINICAL TRIAL: NCT05211804
Title: Mechanisms of Retinal Revascularization and Clinical Indicators of Neovascular AMD Relapse
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21-06505
Record Dates: First submitted 2021-12-16; First posted 2022-01-27 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-03

CONDITIONS: Wet Macular Degeneration
Keywords: age related macular degeneration; age-related macular degeneration; wet age related macular degeneration; wet age-related macular degeneration; Optical Coherence Tomography Angiography; Optical Coherence Tomography; anti vascular endothelial growth factor; neovascular age related macular degeneration; neovascular age-related macular degeneration
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration | interventions — sulphadicramide; aflibercept; Bevacizumab; Ranibizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear film on Schirmers test stored in microtubes at -80°C for biochemical analyses.
  Blood plasma stored in microtubes at -80°C for biochemical analyses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment-naïve: 15 patients not previously receiving anti-VEGF treatment for nAMD.
  Interventions: Drug: Ophthalmic Drugs
- Undergoing treatment: 15 patients already undergoing treatment with anti-VEGF for nAMD.
  Interventions: Drug: Ophthalmic Drugs

INTERVENTIONS:
Drug: Ophthalmic Drugs — Patients will receive the same treatment as if not a part of the project
  Other Names: Aflibercept, Bevacizumab, Ranibizumab

SUMMARY:
Age-related macular degeneration (AMD) is a chronic and progressive eye disease and is one of the leading causes of vision impairment globally. AMD is referred to as either the dry or the wet type, where the wet type (also called neovascular-AMD or nAMD) is a later stage of the disease with neovascularization and retinal edema being the main attributes. This will usually cause subacute distortion or loss of central vision in patients. Since 2004, a successful treatment alternative for nAMD has been ocular injections with anti-VEGF (anti-Vascular Endothelial Growth Factor), causing the neovascularization and edema to regress and vision to improve. However, injections have to be repeated, usually requiring 8 injections or more during the first year of treatment. This can cause both a risk for serious adverse effects and is a significant financial drain on health care resources.

Patients undergoing treatment are at risk for retinal edema recurrence. The time interval tolerated between injections is individual, and the accepted treatment strategy of today is to gradually, in a stepwise manner, increase the interval between injections. For some patients this extension is well tolerated, but for many patients relapse of proliferations and retinal edema will recur. With state-of-the-art technology OCT-A (optical coherence tomography-angiography) in combination with the clinically, well established examination method of OCT (optical coherence tomography), the project group will study the phenotypic vessel and tissue changes that occur in between injections. Furthermore, the investigators will measure cytokines, chemokines and growth factors in blood samples and the tear film during different treatment stages to see if any single factor is prognostic for poorer response to treatment or relapse.

In the short term, the project group hope that the knowledge gained from this project could lead to a better understanding of the mechanisms behind nAMD neovascular relapse and to apply this to routine screening in the clinics. In the longer term, the project group hope that elucidating the physical mechanisms and molecular changes could enable new targeted therapies to be developed.

Aim 1: To characterize the phenotype of vessels in relapsing nAMD patients and compare to those without relapse using OCT-A imaging Aim 2: To investigate retinal edema and choroidal thickness in correlation with neovascular changes of relapsing nAMD Aim 3: To measure cytokines, chemokines and growth factors in the tear film before and during treatment with anti-VEGF for nAMD

With our main hypothesis being: Relapse of nAMD in patients occurs principally through reconfiguration and vasodilatation of persistent non-regressed vessels following anti-VEGF treatment, while fully regressed vessels remain dormant

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be 18 years or older
* Newly diagnosed nAMD (group 1) or nAMD treatment for at least 1 year (group 2), both with typical neovascular findings on OCT-A
* Patients with acceptable travel distance to the hospital
* Patients accepting to be part of the study

Exclusion Criteria:

* Other non-AMD macular disorders
* A spherical equivalent of -6 diopters or less
* Opacities of the visual axis; Changes of the cornea, anterior chamber, lens or vitreous cavity causing image acquisition artefacts
* Patients not able to attend extra controls due to age, illnesses or other factors
* Contraindications of intraocular injection therapy; Active ocular or periocular infection, active and serious intraocular inflammation, hypersensitivity to the drug or recent stroke / heart attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from nAMD patients in the clinic at Eye dep. Sorlandet Hospital Arendal.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Neovascular changes during nAMD relapse assessed by the use of Optical Coherence Tomography Angiography | 12 months after inclusion of patients
  Images gathered from OCTA imaging will be collected and vessel phenotype will be compared between different treatment stages to identify how vessels develop over time. The attributes that will be measured are feeder vessel thickness and to assess if new vessels develop "de novo" or by using old vessel pathways. The investigators intend to describe these findings and there are no planned metric measurements. This outcome is considered a descriptive, qualitative outcome.

SECONDARY OUTCOMES:
Choroidal thickness in nAMD patients undergoing treatment with anti-VEGF will be measured by the use of a caliper tool (metric scale) in the Optical Coherence Tomography software | 12 months after inclusion of patients
  Choroidal thickness will be measured by the use of a caliper tool in the OCTA software and the thickness measured will be compared between different treatment stages of nAMD.
Tear film of nAMD patients at different treatment stages to be collected by Schirmers test and further biochemically analysed | 12 months after inclusion of patients
  Levels of cytokines, chemokines and growth factors will be compared between the different treatment stages of nAMD. This will also be compared to the different levels detected i blood samples done at the same time points. Only for the treatment-naïve group.
Blood samples of nAMD patients at different treatment stages will be collected in microtubes and further biochemically analysed | 12 months after inclusion of patients
  Levels of cytokines, chemokines and growth factors will be compared between the different treatment stages of nAMD. This will also be compared to the different levels detected i tear samples done at the same time points. Only for the treatment-naïve group.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Lagali, Principal Investigator — Sorlandet Hospital HF
Locations (1):
- Sorlandet Hospital HF, Arendal, Agder, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Currently there is not a plan to share individual data outside the project group due to confidentiality. If the investigators later would want to do this, new applications to the correct boards are needed.